CLINICAL TRIAL: NCT06482177
Title: The COAT Trial: Cequa's Onset of Action Trial: an Investigation of CEQUA's Speed of Onset in Improving Ocular Surface Health in Dry Eye Patients
Brief Title: The COAT Trial: Cequa's Onset of Action Trial
Acronym: COAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2303
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dry Eye Disease (Other): Patient with dry eye disease
  Interventions: Drug: Cyclosporine ophthalmic solution

INTERVENTIONS:
Drug: Cyclosporine ophthalmic solution — Cyclosporine BID in the study eye
  Other Names: Cequa

SUMMARY:
Cequa's Onset of Action Trial: an Investigation of CEQUA's Speed of Onset in Improving Ocular Surface Health in Dry Eye Patients

DETAILED DESCRIPTION:
The purpose of this study is to examine the speed of onset of CEQUA ™ in improving the ocular surface among patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

*Patients with the following signs: Central or inferior corneal fluorescein staining defined by the Oxford Scale Reduced tear break up time (TBUT) ≤ 10 seconds.

* Able to comprehend and sign a statement of informed consent.
* Willing and able to complete all required postoperative visits.

Exclusion Criteria:

* Ocular surgery (e.g., intraocular, oculoplastic, corneal, or refractive surgical procedure) performed within the last 3 months or at any time that in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Clinically significant ocular trauma.
* Active ocular Herpes simplex or Herpes Zoster infection
* Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
* Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan, or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
* Active, systemic, or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the study findings.
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis.
* Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
* Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
* Participation in this trial in the same patient's fellow eye
* Patients who are under age 18, pregnant or breastfeeding, or who may become pregnant during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change in corneal high order aberrations (HOA) | After 7, 14, and 28 days of treatment
  Change in corneal HOA

SECONDARY OUTCOMES:
Change in corneal staining | After 7, 14, 28 days of treatment
  Corneal staining

OTHER OUTCOMES:
Change in best corrected visual acuity | After 7, 14, and 28 days of treatment
  Best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Harvard Eye Associates
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States